CLINICAL TRIAL: NCT00522964
Title: Educational Intervention on Weight Management in Chinese American Children
Brief Title: Educational Intervention on Weight Management in Chinese-American Children
Acronym: ABC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Jyu-Lin Chen; Assistant Professor, UCSF
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: KL2RR024130 (NIH); NIH KL2 RR024130
Record Dates: First submitted 2007-08-28; First posted 2007-08-30 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Overweight
Keywords: Chinese-American; Children; Obesity; health behaviors; Behavioral intervention; normal
MeSH Terms: conditions — Overweight; Obesity; Health Behavior | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental)
  Interventions: Behavioral: behavioral intervention

INTERVENTIONS:
Behavioral: behavioral intervention — The intervention is based on Social Cognitive Theory and principles of Chinese culture and practices. The intervention program includes a one-hour small-group session for eight weeks for children and two 2-hour small-group sessions for parents.

SUMMARY:
A randomized study is proposed to determine effects of 8 weeks of an interactive multimedia educational program compared to waiting list control group on improving health and weight status in Chinese-American children, ages 8 and 10, over a 6 months period. A total of 60 Chinese-American children and their families will be randomized to either the intervention group or waiting list control group. The intervention is based on Social Cognitive Theory and principles of Chinese culture and practices. The intervention program includes a one-hour small-group session for eight weeks for children and two 2-hour small-group sessions for parents. Baseline data will be collected before assigning the children to the intervention or control group. Follow-up data will be collected immediately after the intervention and 3 months and 6-months post intervention. A repeated measures (longitudinal) design employing a linear mixed models approach will be used for analysis.

DETAILED DESCRIPTION:
The most recent data indicate that the prevalence of overweight and risk of becoming overweight among Chinese Americans aged 6 to 11 years is 31%. Several physical and psychosocial health consequences are associated with childhood overweight and poor physical fitness, including cardiovascular diseases (CVDs), sleep disorders, type 2 diabetes mellitus, low self-esteem, and social withdrawal. Chinese Americans are at a higher risk of developing CVDs and T2DM than are non-Hispanic whites possibly due to genetic differences in body composition and metabolic responses. Therefore, developing programs that focus on preventing overweight and promoting healthy lifestyles in early childhood is imperative in preventing long-term adverse effects of overweight, especially in Chinese-Americans. A randomized study is proposed to examine feasibility and efficacy of a child-centered and family-focused behavioral intervention on improving health behavior, psychosocial function, anthropometrics, and biochemical indices in Chinese-American children.

The primary aim is to test the effect of a multimedia behavioral intervention on the health behaviors, psychosocial function, and anthropometrics of Chinese-American children, ages 8 and 10.

Aim 1a. Children in the intervention group will report a healthier dietary intake (more vegetable and fiber and lower fat) than will children in the control group at 2 months, 4 months and 6-months post baseline assessment.

Aim 1b. Children in the intervention group will report being more active than will children in the control group at 2 months, 4 months and 6-months post baseline assessment.

Aim 1c. Children in the intervention group will report a significantly higher self-efficacy in relation to nutrition and physical activity than will children in the control group at 2 months, 4 months and 6-months post baseline assessment.

Aim 1d. Children in the intervention group will report significantly better coping than will children in the control group at 2 months, 4 months and 6-months post baseline assessment.

Aim 1e. Children in the intervention group will report a greater decrease in BMI than will children in the control group at 6-months post baseline assessment.

Aim 1f. Children in the intervention group will experience a greater decrease in fat mass than will children in the control group at 6-months post baseline assessment.

The secondary aim is to examine the effect of the multimedia behavioral intervention on biochemical indices of health in Chinese-American children, ages 8 and 10.

Aim 2a. Children in the intervention group will experience an increase in insulin sensitivity vs. children in the control group at 6-months post baseline assessment.

Aim 2b. Children in the intervention group will experience an improvement in cholesterol, high-density lipoproteins (HDLs), low-density lipoproteins (LDLs), and triglycerides (TGs) vs. children in the control group at 6- months post baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

Eight and ten-year-old Chinese-American children and their parents will be eligible for enrollment if they meet the following criteria:

* Children must be overweight (BMI is between 85th% tile and 94th% tile) or obese (BMI is greater than 95th% tile) based on CDC growth chart
* The adult and child self-identify ethnicity to be Chinese or of Chinese origin and they must reside in the same household to be eligible. A dyad of one adult and one child is the minimum necessary for a household to participate. Two adults per child will be encouraged to participate.
* The child is able to speak and read English.
* The child is in good health, defined as free of an acute or life-threatening disease and able to attend to activities of daily living such as going to school.
* Parents are able to speak English, Mandarin, or Cantonese, and are able to read in English or Chinese and to complete questionnaires.

Exclusion Criteria:

* Children with chronic health problems that include any dietary modifications or activity limitations will be excluded (e.g., diabetes, exercise-induced asthma).

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
health behaviors, psychosocial function, and anthropometrics of Chinese-American children | 6 months

SECONDARY OUTCOMES:
insulin, cholesterol, high-density lipoproteins (HDLs), low-density lipoproteins (LDLs), and triglycerides (TGs) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jyu-Lin Chen, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States